

## **Clinical Trial**

# **PROTECTUP**

## **Protocol**

<u>P</u>hysiological vs <u>R</u>ight ventricular pacing <u>O</u>utcome <u>T</u>rial <u>E</u>valuated for Brady<u>C</u>ardia <u>T</u>reatment <u>Upg</u>rades

Version 5.0

**SPONSOR:** Imperial College London

FUNDER: Academic grant Heart Research UK

TRIAL COORDINATION CENTRE: Hammersmith Hospital London

NRES reference: NRES Committee Greater Manchester West

Clinicaltrials.gov reference: NCT06052475

#### Protocol authorised by:

| Name & Role | Date | Signature |
|-------------------|------|-----------|
| Daniel Keene (CI) | | |

## **Trial Management Group**

| Chief Investigator | Dr. Daniel Keene |
|--------------------|--------------------------|
| Co-investigators: | Dr Nandita Kaza |
| | Dr. Matthew Shun-Shin |
| | Dr. Zachary Whinnett |
| | Professor Darrel Francis |
| Statistician | Professor Darrel Francis |
| Trial Manager | Miss Aya Khalil |

Ref: 23HH8156

IRAS ID: 323165 V5 – 29-07-2024

Clinical Queries

Clinical queries should be directed to Dr Daniel Keene (d.keene@imperial.ac.uk)

**Sponsor** 

Imperial College London is the main research Sponsor for this Trial. For further information regarding

the sponsorship conditions, please contact the Head of Regulatory Compliance at:

Research Governance and Integrity Team

Imperial College London and Imperial College Healthcare NHS Trust

Room 215, Level 2, Medical School Building

Norfolk Place

London, W2 1PG

Tel: 0207 594 1862

Imperial College - Research Governance and Integrity Team (RGIT) Website

**Funder** 

This Trial is funded by an academic grant from Heart Research UK.

This protocol describes the Trial ('Physiological vs Right ventricular pacing Outcome Trial Evaluated for bradyCardia Treatment Upgrades IRAS ID 323165) and provides information about procedures for entering participants. Every care was taken in its drafting, but corrections or amendments may be necessary. These will be circulated to investigators in the trial. Problems relating to this trial should be

referred to the Chief Investigator in the first instance.

This trial will adhere to the principles outlined in the NHS Research Governance Framework for Health

and Social Care (2nd edition).

It will be conducted in compliance with the protocol, the Data Protection Act and other regulatory

requirements as appropriate.

## **Table of Contents:**

| 1.1 | BACKGROUND AND RATIONALE FOR CURRENT TRIAL | 6 |
|-----------|--------------------------------------------|----|
| 2. TF | RIAL OBJECTIVES | 7 |
| 3. TF | RIAL DESIGN | 8 |
| 4. | PARTICIPANT ENTRY | 10 |
| 4.1 | PRE-REGISTRATION EVALUATIONS | 10 |
| 4.2 | INCLUSION CRITERIA | 10 |
| 4.3 | EXCLUSION CRITERIA | 10 |
| <i>5.</i> | ADVERSE EVENTS | 10 |
| 5.1 | DEFINITIONS | 10 |
| 5.2 | REPORTING PROCEDURES | 11 |
| <i>6.</i> | ASSESSMENT AND FOLLOW UP | 12 |
| <i>7.</i> | STATISTICS AND DATA ANALYSIS | 13 |
| 8. | REGULATORY ISSUES | 14 |
| 8.1 | ETHICS APPROVAL | 14 |
| 8.2 | CONSENT | 14 |
| 8.3 | CONFIDENTIALITY | 15 |
| 8.4 | INDEMNITY | 15 |
| 8.5 | SPONSOR | 15 |
| 8.6 | FUNDING | 15 |
| 8.7 | AUDITS | 16 |
| 9. | TRIAL MANAGEMENT | 16 |
| 10 | PUBLICATION POLICY | 16 |



## **TRIAL SUMMARY**

| TITLE | Physiological vs Right ventricular pacing Outcome Trial Evaluated for brady Cardia Treatment Upgrades |
|---|---|
| DESIGN | It is a double-blind, randomized multi-centre trial. A total of 155 participants, considered for clinical pacemaker upgrade (placement of an additional pacing lead aiming to deliver more physiological ventricular activation; either within the coronary sinus (biventricular pacing) or at the Bundle of His or Left Bundle Area (Conduction System Pacing) undergo randomised crossover periods of 1 month and 6 months in either RV pacing (continued original pacing strategy) or with the more physiological pacing strategy. The crossover periods will enable assessment of the utility of clinically performed device upgrades. |
| AIMS | This trial will aim to study the utility of upgrading patients to physiological pacing from right ventricular (RV) pacing focusing on patients with mild or moderate impairment of cardiac function. |
| OUTCOME<br>MEASURES | The primary outcome measure will be SF36 quality of life questionnaire physical component summary score |
| POPULATION | The trial will recruit 155 participants scheduled for clinical device upgrade either at the time of generator replacement or at any other timepoint. |
| ELIGIBILITY | Adults with an LVEF 35-50% AND >40% RV pacing AND at least one of the following: (1) EF reduced by >5% or increase in LVESV by 10ml since implant (2) NT-proBNP >250ng/L in sinus rhythm (3) NT-proBNP >750ng/L in Atrial Fibrillation (4) Left Atrial Volume index >30ml/m² (5) Regular loop diuretics prescribed (6) Decline in daily patient activity by >1hour per day since implant (7) Decrease in device measured thoracic impedance (8) Patient reported decline in functional class / exercise tolerance |
| DURATION | <ul> <li>18 months for patient recruitment</li> <li>15 month follow up period.</li> <li>3-month analysis and provisional reporting</li> <li>Total duration: 36 months</li> </ul> |

Ref: 23HH8156

IRAS ID: 323165 V5 - 29-07-2024

© Imperial College of Science, Technology and Medicine



#### **GLOSSARY OF ABBREVIATIONS**

AE Adverse Event

AR Adverse Reaction

CA Competent Authority

CCMO Central Committee on Research Involving Human Subjects

DSMB Data Safety Monitoring Board

EU European Union

EudraCT European drug regulatory affairs Clinical Trials

GCP Good Clinical Practice

GDPR General Data Protection Regulation

HFrEF Heart Failure with reduced Ejection Fraction

IB Investigator's Brochure

IC Informed Consent

IMP Investigational Medicinal Product

IMPD Investigational Medicinal Product Dossier

LVEF Left Ventricular Ejection Fraction

LBB Left Bundle Branch

LBBB Left Bundle Branch Block
LBBP Left Bundle Branch Pacing

NYHA New York Heart Association functional class

(S)AE (Serious) Adverse Event

Sponsor The sponsor is the party that commissions the organisation or performance of

the research, for example a pharmaceutical

company, academic hospital, scientific organisation or investigator. A party that provides funding for a trial but does not commission it is not regarded as the

sponsor but referred to as a subsidising party.

SUSAR Suspected Unexpected Serious Adverse Reaction

#### **KEYWORDS**

Cardiac Resynchronisation

**HIS Bundle Pacing** 

Left Bundle Branch Pacing

**Device Upgrade** 

Ref: 23HH8156

IRAS ID: 323165 V5 – 29-07-2024

1. INTRODUCTION

1.1 BACKGROUND AND RATIONALE FOR CURRENT TRIAL

Today, patients who are scheduled to receive a pacemaker for the first time and are expected

to have high burden of RV pacing (>20/40%), with any (i. e., mild, moderate, or severe) degree

of LV impairment are guideline recommended to receive a physiological pacing strategy rather

than RV pacing. RCTs, observational studies and meta-analysis data provide strong evidence

that this improves patient symptoms, echocardiographic markers, morbidity and even

mortality.

Patients with existing RV pacemakers, are frequently upgraded clinically using this same

rationale, existing observational data sets and meta-analysis data that physiological pacing

strategies are less damaging to cardiac function than ongoing RV pacing. RCTs currently

though have only evaluated upgrade procedures in patients with severe LV impairment.

The trial aims to provide high-quality RCT evidence for upgrading patients to physiological

pacing strategies for those patients with mild or moderate LV impairment. This represents a

large patient cohort susceptible to morbidity and mortality from continued RV pacing. RV

pacing saves lives in the short-term by preventing bradycardia but can lead to LV impairment

in the longer term, increasing rates of heart failure and death. Two RCTs have demonstrated

the harm of RV pacing.

In the DAVID trial, patients with an impaired LV were randomised to back-up pacing

(minimising RV pacing), or obligatory RV pacing (maximising RV pacing). The group that

received a high percentage of RV pacing had markedly higher rates of heart failure and death

from 16.1% to 26.7% (HR 1.61). We have previously a meta-analysis of randomized controlled

trials (RCTs) and observational studies assessing device upgrades. We analysed studies of

biventricular (BiV) pacing (6 RCTs of 161 patients, and 46 observational studies of 2,795

patients) and Conduction system pacing (CSP) upgrades (7 studies of 197 patients)

separately.11-68 RCTs of BiV pacing upgrade showed LVEF improvement of +8.4% from

34.4%, and observational studies showed LVEF improvement of +8.5% from 25.7%.

Observational studies of CSP upgrade showed LVEF improvement of +11.2% from 38.4%.

LVESV decreased significantly by -25.4mls, -23.7mls, and -19.8mls in BiV RCTs, BiV

observational studies and CSP observational studies respectively. NYHA class improved by -

0.4, -0.8 and -1.0 respectively. RCTs of BiV pacing upgrade found improvements in Minnesota

Heart Failure Score (-6.9 points) and peak oxygen uptake (+1.1ml/kg/min,). This was also

seen in observational BiV upgrade studies (-19.7 points and +2.6ml/kg/min respectively).

2. TRIAL OBJECTIVES

We aim to test whether the positive effects of upgrading to physiological pacing strategies

translate into benefit for patients with mild, or moderate impairment to their ventricles as a

result of RV pacing.

We hypothesise that upgrade to physiological pacing strategies even when the extent of

cardiac impairment is only mild or moderate will result in significant symptomatic and

physiological benefit.

**Primary Objectives:** 

This trial will evaluate, in patients with existing RV pacemakers and only mild or

moderate LV impairment, whether clinically used modern physiological pacing

strategies rather than continued RV pacing improve quality-of-life as measured by SF-

36 questionnaire physical component summary score under double-blinded

conditions?

**Secondary Objectives:** 

1. In patients with RV pacemakers and existing mild to moderate LV impairment, what is

the effect of modern physiological pacing strategies rather than continued RV pacing

on:

(a) Left ventricular ejection fraction.

(b) Left ventricular end systolic index.

(c) Quality of life questionnaires as measured by the Minnesota Living with Heart

Failure Questionnaire, EQ5D5L and SF-36 questionnaire overall score.

(d) Six-minute walk test

(e) Atrial fibrillation

(f) Patient preference based on blinded symptomatic preference

2. Is upgrading to physiological pacing more beneficial at time of generator change or at

an earlier timepoint?

3. What are the complications associated with upgrade procedures?

3. TRIAL DESIGN

3.1 Trial protocol

Eligible patients will be those considered clinically for a device upgrade by their clinical team.

Patients will be invited to participate in the trial before their planned clinical procedure.

All participants will undergo an upgrade procedure and receive either Conduction System

Pacing (His or Left Bundle pacing) as first line approach or Biventricular Pacing if Conduction

System Pacing cannot be delivered. An experienced operator will carry out the procedures.

Participants will be allocated in blinded random fashion to pacing periods using randomisation

software (sealed envelope). They will be randomised to either having their 'physiological

pacing strategy active OR continued RV pacing. Participants will undergo two one-month

crossover periods and then two six-month crossover periods. Participants undergo the same

evaluations at each visit.

At baseline and at the end of each period the participants will have the following assessed:

Validated Quality-of-Life Questionnaire SF-36 questionnaire

Minnesota Living with Heart Failure

- EQ5D5L questionnaires.

6-min walking test

blood tests including NT-proBNP

Echocardiography

- data collection regarding any heart failure hospitalisations

medication list

Pacing parameters: arrhythmia burden, pacing percentages, daily patient activity.

After the 2x 1-month periods and after the 2x 6-month periods, blinded patient preference will

be asked on a 7-point preference scale. Again, at the end, they will be asked for their

symptomatic preference. Participants will be invited to participate in the trial before their

planned clinical investigation. Each participant will have a run-in period of 1 month, and then

be followed-up at one-monthly intervals by a central trial hub followed by six-monthly intervals.

3.2 Trial End

The trial ends when the last enrolled trial participant completes their last follow-up at fifteen

months following their upgrade date. The trial end date is defined as the date the last

participant's second 6-month period comes to an end and all the research procedures

occurring at this timepoint are completed.

Any procedures occurring as part of the research study will be reviewed in the Imperial College

Healthcare NHS Trust weekly multi-disciplinary team meeting, which includes a group of

consultant cardiologists. Any complications resulting from these research procedures will be

formally presented, evaluated and discussed within the MDT. If any concerning trends are

identified as a result of these research procedures, a decision will be made to end the trial

early.

3.3 Trial outcome measures

Primary outcome measure:

The primary outcome is quality-of-life as measured by SF-36 questionnaire physical

component summary score under double-blinded conditions. It is mandatory for participants

to complete the SF-36 questionnaire physical component summary score at baseline, months

1, 2, 8, and 14 for essential data points. Additional submissions between these periods are

optional, providing participants flexibility for more frequent updates on their quality of life.

Secondary outcome measure:

1. In patients with RV pacemakers and existing mild to moderate LV impairment, what is

the effect of modern physiological pacing strategies rather than continued RV pacing

on:

(a) Left ventricular ejection fraction.

(b) Left ventricular end systolic index.

(c) Quality of life questionnaires as measured by the Minnesota Living with Heart

Failure Questionnaire, EQ5D5L and SF-36 questionnaire overall score.

(d) Six-minute walk test

(e) Atrial fibrillation

(f) Patient preference based on blinded symptomatic preference.

2. Is upgrading to physiological pacing more beneficial at time of generator change or at

an earlier timepoint?

3. What are the complications associated with upgrade procedures?

4. PARTICIPANT ENTRY

4.1 PRE-REGISTRATION EVALUATIONS

We will recruit patients who are referred for clinically indicated cardiac resynchronisation

therapy upgrade.

PIC sites will identify patients meeting eligibility criteria with high burden RV pacing who are

clinically indicated for an upgrade procedure. These patients will then undergo their upgrade

procedure at ICHT - Hammersmith Hospital (as these PIC sites do not offer the conduction

system pacing upgrade procedure).

4.2 INCLUSION CRITERIA

Adults with an RV pacemaker and LVEF 35-50% who are clinically indicated for an upgrade

procedure plus any of the following:

o EF reduced by >5% or increase in LVESV by 10ml since implant.

NT-proBNP >250ng/L in sinus rhythm

NT-pro BNP>750ng/L if AF

Left atrial volume index >30 mL/m²

Regular loop diuretics prescribed.

Decline in daily patient activity by >1 hour per day since implant.

o Decrease in device measured thoracic impedance.

o Patient reported decline in functional class / exercise tolerance.

4.3 EXCLUSION CRITERIA

Inability to provide informed consent.

o Aged under 18

o Pregnant women.

5. ADVERSE EVENTS

Any complications resulting from these research procedures will be formally presented,

evaluated and discussed within the Imperial College Healthcare NHS Cardiology MDT. If any

concerning trends are identified as a result of these research, a decision will be made to end

the trial early.

5.1 **DEFINITIONS** 

Adverse Event (AE): any untoward medical occurrence in a patient or clinical trial subject.

Serious Adverse Event (SAE): any untoward and unexpected medical occurrence or effect

that:

Results in death

o Is life-threatening – refers to an event in which the subject was at risk of death at the

time of the event; it does not refer to an event which hypothetically might have caused

death if it were more severe.

o **Requires hospitalisation**, or prolongation of existing inpatients' hospitalisation.

Results in persistent or significant disability or incapacity

Is a congenital anomaly or birth defect.

Medical judgement should be exercised in deciding whether an AE is serious in other

situations. Important AEs that are not immediately life-threatening or do not result in death or

hospitalisation but may jeopardise the subject or require intervention to prevent one of the

other outcomes listed in the definition above should also be considered serious.

5.2 REPORTING PROCEDURES

All adverse events should be reported. Depending on the nature of the event, the reporting

procedures below should be followed. Any questions concerning adverse event reporting

should be directed to the Chief Investigator in the first instance.

5.2.1 Non-serious AEs

All such events, whether expected or not, should be recorded.

5.2.2 Serious AEs

An SAE form should be completed and emailed to the Chief Investigator within 24

hours. However, relapse and death due to pre-existing medical problems and

hospitalisations for elective treatment of a pre-existing condition do not need reporting

as SAEs.

All SAEs should be reported to the REC (NRES Committee Greater Manchester West)

where in the opinion of the Chief Investigator, the event was:

'related', i.e., resulted from the administration of any of the research

procedures; and

o 'unexpected', i.e., an event that is not listed in the protocol as an expected

occurrence.

Reports of related and unexpected SAEs should be submitted within 15 days of the Chief Investigator becoming aware of the event, using the NRES SAE form for non-

IMP studies. The Chief Investigator must notify the Sponsor of all related and

unexpected SAEs.

Local investigators should report any SAEs as required by their Local Research Ethics

Committee, Sponsor and/or Research & Development Office.

**Contact details for reporting SAEs:** 

RGIT@imperial.ac.uk

Please send SAE forms to: d.keene@imperial.ac.uk

Tel: 020 7594 1093 (Mon to Fri 09.00 – 17.00)

6. ASSESSMENT AND FOLLOW UP

Post-procedure, the participant will be followed up by their clinical team. Pacing checks will be

undertaken as per clinical protocol and standard of care. All patients pacing notes will be

marked as indicating the patient is involved in a clinical trial and clinical team should not

disclose to the patient the pacing period allocation.

At every timepoint for research follow-ups following the participant's pacemaker upgrade i.e.

at the 1-month, 2-months, 8-months and 14-month timepoint – we will collect:

o Validated Quality-of-Life Questionnaire SF-36, Minnesota Living with Heart Failure,

and EQ5D5L questionnaires.

6-min walking test

blood tests incl. NT-proBNP

Echocardiography

data collection regarding any heart failure hospitalisations

medication list

o Pacing parameters: arrhythmia burden, pacing percentages, daily patient activity.

Patient's Quality of life will be assessed monthly via the SF36 validated quality of life

questionnaire and this will be done either electronically or via telephone, according to patient's

preference. Patient symptoms will also be assessed monthly via custom symptom

questionnaires (non-validated) in the one-month crossover periods and then monthly in the

six-month crossover periods. Participants can choose whether to participate in monthly

questionnaires, and it's entirely optional for those who are willing to take part in the monthly

assessment.

Incidental findings identified as part of the research protocol will be reviewed and reported by

trained clinical members of the research team. Any incidental findings identified will be

communicated to the participant's clinical team as well as their GP as per standard protocol.

7. STATISTICS AND DATA ANALYSIS

7.1 Sample size calculations:

The sample size calculation for the PROTECT UP cross over RCT is as follows:

Assuming standard deviation of difference of sequential measurements of SF35 of 10 units,

136 patients (68 in each arm - on/off or off/on) would provide 80% power at the 5%

significance threshold to detect a 3.5-unit difference in SF36 Physical Component Score

between the upgraded physiological pacing strategy and standard of care RV pacing. To

account to loss to follow-up of 12% we will recruit and randomise 155 patients. Patients will

only be randomised after successful upgrade.

Our primary outcome will use the longest available comparable period, ideally the 6-month

duration periods, but if participants have elected to withdraw because of overwhelming patient

perceived blinded benefit/harm we will use their blinded QOL assessment from the longest

available period. If participants wish to withdraw during a pacing period because of poor

symptoms we will aim to perform endpoint assessment at that point in a blinded fashion and

use that data.

7.2 Statistical Analysis:

Analysis will be performed according to the ITT principle and all statistical tests will be two-

tailed with a 5% significance level.

The primary and secondary continuous secondary endpoints (SF-36 individual and global

components, MLWHF, daily patient activity, LVEF, LVESI, 6-minute walk test and patient

preference, BNP) will be analysed using a mixed-effect modelling approach, including the

treatment and randomisation order as independent variables.

For time-to-event endpoints (death and hospitalisation for heart failure), the hazard ratio and

respective 95% confidence interval will be computed using the Cox proportional hazards

regression model, or appropriate alternative.

In secondary analysis the model will be adjusted for clinical important confounders that will be

pre-specified in the statistical analysis plan. The underlying assumptions of any fitted model

will be assessed as appropriate.

We will test the impact of relevant subgroups (time of upgrade (ERI vs Early upgrade), timing

of improvement (one month vs 6 month) presence of AF, percentage pacing, BIV vs CSP

pacing approach) by testing the interaction of these variables on the treatment.

Data and all appropriate documentation will be stored for a minimum of 10 years after the

completion of the trial, including the follow-up period.

8. REGULATORY ISSUES

8.1 ETHICS APPROVAL

The Trial Coordination Centre has obtained approval from the Greater Manchester

West Research Ethics Committee (REC) and Health Research Authority (HRA). The

trial must also receive confirmation of capacity and capability from each participating

NHS Trust before accepting participants into the trial, or any research activity is carried

out. The trial will be conducted per the recommendations for physicians involved in

research on human subjects adopted by the 18th World Medical Assembly, Helsinki

1964 and later revisions.

8.2 CONSENT

Consent to enter the trial must be sought from each participant only after a complete

explanation, an information leaflet offered, and time allowed for consideration. Signed

participant consent should be obtained. There will be no pre-specified window for

consenting patients; patients can consent to take part in the trial up until the day of

their procedure. The right of the participant to refuse to participate without giving

reasons must be respected.

Patient consent for a referral to the research team and transfer of their data will be

documented in patient notes.

After the participant has entered the trial, the clinician remains free to give alternative

treatment to that specified in the protocol at any stage if they feel it is in the participant's

best interest. Still, the reasons for doing so should be recorded. In these cases, the

participants remain within the trial for follow-up and data analysis. All participants are

free to withdraw from the protocol treatment at any time without giving reasons or

prejudicing further treatment

8.3 CONFIDENTIALITY

The Chief Investigator will preserve the confidentiality of participants participating in

the trial and is registered under the Data Protection Act.

Data will be pseudonymised using a number code which can only be linked to

personally identifiable information kept in a separate record. The code will replace all

personally identifiable information in the primary records used for the trial.

8.4 INDEMNITY

Imperial College London holds negligent harm and non-negligent harm insurance

policies, which apply to this trial.

8.5 SPONSOR

Imperial College London will act as the main Sponsor for this trial. Delegated

responsibilities will be assigned to the NHS trusts taking part in this trial.

8.6 FUNDING

The Trial is funded by an academic grant from the Heart Research UK Charity.

As we are requiring participants to attend hospital for reasons aside from their usual

clinical care, we will be able to offer expenses for participant's travel and refreshments.

All the trial visits will be undertaken at Imperial College London, Hammersmith

Hospital. Neither the clinical team nor members of the research team will receive any

financial incentives as a result of inviting participants to take part in this research.

8.7 AUDITS

The trial may be subject to inspection and audit by Imperial College London under their

remit as the sponsor and other regulatory bodies to ensure adherence to GCP and the

NHS Research Governance Framework for Health and Social Care (2<sup>nd</sup> edition).

An independent Data Monitoring Committee (DMC) will be set up to review data for

safety and efficacy at regular intervals. The DMC will prepare a charter (in line with the

DAMOCLES recommendations) outlining their responsibilities and reporting

requirements.

An independent Data Monitoring Committee (DMC) will be set up to review data for

safety and efficacy at regular intervals. The DMC will prepare a charter (in line with the

DAMOCLES recommendations) outlining their responsibilities and reporting

requirements.

9. TRIAL MANAGEMENT

The day-to-day management of the trial will be coordinated through Dr Daniel Keene

(d.keene@imperial.ac.uk), Dr Nandita Kaza (n.kaza@imperial.ac.uk) and Aya Khalil

(akhalil@ic.ac.uk).

10. PUBLICATION POLICY

We will seek to publish the trial's results in internal reports, scientific presentations and peer-

reviewed scientific journals. The scientific team will make all analyses and decisions to publish

and will not be influenced by the funder.